CLINICAL TRIAL: NCT06831864
Title: Heart Failure With Reduced Ejection Fraction Polypill Implementation Strategy in Sri Lanka: A Pilot Randomized Trial
Brief Title: Heart Failure With Reduced Ejection Fraction Polypill Implementation Strategy in Sri Lanka
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: The George Institute (Other); RemediumOne (Unknown); Centre for Chronic Disease Control, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202306038
Record Dates: First submitted 2024-04-10; First posted 2025-02-18 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: HFrEF; Heart Failure; Heart Failure with Reduced Ejection Fraction; Sri Lanka; Polypill
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparator (control) arm (Other): Participants in the comparator control arm will receive usual care, as per their physician's discretion.
  Interventions: Other: Comparator Arm
- Study Intervention arm (Experimental): Participants in the intervention group will be provided the HFrEF polypill by the study.
  Interventions: Drug: HFrEF Polypill

INTERVENTIONS:
Drug: HFrEF Polypill — The heart failure with reduced ejection fraction (HFrEF) polypill will include 4 guideline recommended medications used to treat HFrEF patients. The dose of initiation and titration will be at the investigator's discretion.
  HFrEF polypill strength 1: bisoprolol 2.5 mg + losartan 25 mg + eplerenone 25 mg + dapagliflozin 10 mg; HFrEF polypill strength 2: bisoprolol 5 mg + losartan 50 mg + eplerenone 25 mg + dapagliflozin 10 mg; HFrEF polypill strength 3: bisoprolol 10 mg + losartan 100 + eplerenone 50 mg + dapagliflozin 10 mg
  Arms: Study Intervention arm
Other: Comparator Arm — Participants in the comparator control group will receive usual care by their healthcare providers. Providers will be encouraged to treat all participants according to international and local clinical practice guidelines.
  Arms: Comparator (control) arm

SUMMARY:
The primary objective of this trial is to see if the research team can successfully recruit participants and carry out study related procedures in Sri Lanka. This will help the research team plan and execute a future large-scale trial in Sri Lanka.

The secondary objective is to assess whether a polypill for patients with heart failure with reduced ejection fraction (a type of heart condition) may help patients adhere to medications without an increase in serious adverse events.

An exploratory objective is to understand the process of implementation.

Participants will be randomly assigned to one of two groups, intervention or usual care. The intervention group will be given four guideline-recommended medications for heart failure with reduced ejection fraction, combined in one over-encapsulated pill, with three dose strength options (at the discretion of their treating physician). Both groups will be observed over 4-weeks of follow-up to assess their medication adherence, clinical symptoms, laboratory measures, health related quality of life, and need for medication adjustment amongst other measures.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥18 years old)
* Diagnosis of heart failure with reduced ejection fraction (HFrEF) including clinical symptoms or clinical signs or natriuretic peptide elevation AND echocardiographic or other evidence of reduced ejection fraction (EF 40%)
* New York Heart Association Class II, III, or IV symptoms

Exclusion Criteria:

* Known contraindication to any of the HFrEF polypill components (e.g., advanced renal disease, bradycardia, allergy, amongst others).
* Significant renal impairment (estimated glomerular filtration rate <=30 mL/min/1.73 m2 or creatinine clearance <=30mL/min).
* Raised serum potassium >5 mEq/L.
* Symptomatic hypotension or systolic BP <100 mmHg as per the average of last 2 of the 3 measurements at visit 1.
* Symptomatic bradycardia or second or third-degree heart block without a pacemaker on ECG review at visit 1.
* Cardiogenic shock and/or current use of inotropes.
* Myocardial infarction, unstable angina, stroke or transient ischemic attack (TIA) within 12 weeks prior to enrollment.
* Women who are pregnant, breastfeeding or of childbearing potential and are not using and do not plan to continue using medically acceptable form of contraception throughout the study (pharmacological or barrier methods).
* Concomitant illness, physical impairment or mental condition which in the opinion of the study team / primary physician could interfere with the conduct of the study including outcome assessment.
* Participation in a concurrent interventional medical investigation or pharmacologic clinical trial. Patients in observational, natural history or epidemiological studies not involving an intervention are eligible.
* Participant's responsible physician believes it is not appropriate for participant to participate in the study.
* Inability or unwillingness to provide written informed consent.
* Involvement in the planning and/or conduct of the study.
* Unable to complete study procedures and/or plan to move out of the study site area in the next 2 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment | 0 - 10 weeks, start of enrollment to completion of participant enrollment
  Feasibility of recruitment based on completion of the following: recruitment of up to 40 participants at a rate of 4 participants per week.
Adherence to study procedures | 0 - 14 weeks, baseline to study end
  Adherence to study procedures based on completion of the following: completion of study-related procedures (screening, randomization, study drug allocation, follow-up procedures, retention, and outpatient transition).

SECONDARY OUTCOMES:
Adherence to overall and individual components of GDMT | 4 weeks
  The secondary outcome is the proportion of individuals with adherence to overall and individual components of GDMT (ACE-I or ARB or ARNi, BB, MRA, and SGLT2i use at any dose in the absence of contraindications) at 4 weeks measured by 1) pill count, and 2) the self-report tool Medication Adherence Report Scale (MARS-5).
Withdrawals due to Adverse Events | From enrollment to the end of treatment at 4 weeks
  Proportion of withdrawals due to adverse events.
Serious Adverse Events | From enrollment to the end of treatment at 4 weeks
  Proportion of participants with any serious adverse events (SAEs) according to the Good Clinical Practice (GCP) definition.
Adverse Events of Special Interest | From enrollment to the end of treatment at 4 weeks
  Proportion of participants with adverse events of special interest (diabetic ketoacidosis, volume depletion [hypotension, syncope, orthostatic hypotension or dehydration all defined clinically], severe hypoglycemic event, lower limb amputation, hyperkalemia, worsening renal function)
Mean Change in Serum Potassium | 4 weeks
  Mean change (from baseline) in continuous serum potassium, controlling for baseline value.
Change in Serum Creatinine | 4 weeks
  Mean change (from baseline) in serum creatinine, controlling for baseline value.

CONTACTS AND LOCATIONS:
Locations (2):
- Sri Lanka (2):
  - National Hospital of Sri Lanka, Colombo
  - Colombo South Teaching Hospital, Colombo

IPD SHARING:
Plan to Share IPD: No
When the study is over, research findings will be available at www.ClinicalTrials.gov and Sri Lanka Clinical Trials Registry. Laboratory results will be shared with participants and their health care providers. The research findings will also be published in the form of research articles or presented at scientific meetings.

REFERENCES:
- [Derived] Agarwal A, de Silva A, Agarwal M, Ajanthan S, Dahanayaka A, Dhurjati R, Fernando C, Galappatthy G, Goss CW, Hively A, Jayagopal PB, Mohanan PP, Patel A, Prabhakaran D, Rahuman M, Rodgers A, Roberts K, Salwa H, Huffman MD, Salam A. Heart failure with reduced ejection fraction polypill implementation strategy in Sri Lanka: design and protocol of a pilot type I hybrid randomised clinical trial. BMJ Open. 2025 Jul 15;15(7):e100952. doi: 10.1136/bmjopen-2025-100952. PMID 40664424
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/33211084/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/34612082/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/37334398/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/39817063/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/39219851/